CLINICAL TRIAL: NCT02285348
Title: Oxidative Stress, Low Grade Inflammation, Tissue Breakdown and Biomarkers in Cerebrospinal Fluid of Patients With Ataxia Telangiectasia
Brief Title: Oxidative Stress, Low Grade Inflammation, Tissue Breakdown and Biomarkers in Cerebrospinal Fluid of A-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Stefan Zielen, Prof. Dr., Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FRA-AT.CSF.2012
Record Dates: First submitted 2014-10-28; First posted 2014-11-07 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Telangiectasia; cerebrospinal fluid; inflammation; proteomic analysis
MeSH Terms: conditions — Ataxia Telangiectasia; Inflammation | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ataxia Telangiectasia (Other): 20 patients with clinically and/or genetically diagnosed Ataxia telangiectasia will get a lumbar puncture
  Interventions: Procedure: Lumbar puncture
- Healthy Control (Other): 20 patients without inflammation, infection or any other pathology of the CNS, in that a lumbar puncture is indicated for either diagnostic or therapeutic reason (i.e. for the exclusion of a meningitis, subarachnoid hemorrhage or in therapeutic liquor drain in idiopathic intracranial hypertension)
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — Lumbar puncture is done according to general practice

SUMMARY:
Ataxia telangiectasia (A-T) is a rare devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability, and cancer susceptibility. The underlying mechanism and process of neurodegeneration leading to loss of cerebellar neurons and neurological function is largely unknown. Laboratory diagnostic approaches to neurodegeneration in A-T are hampered by sampling issues. It is dangerous, impractical, and not ethically to directly sample brain tissue by surgical biopsy. In contrast cerebrospinal fluid (CSF), a fluid that is in direct contact with brain tissue, is relatively easy to sample in a safe procedure (lumbar puncture). The aim of the proposal is to investigate oxidative stress, low grade inflammation and tissue break down in the brain of A-T patients by analyzing CSF. In addition the alterations in protein expression related to A-T will be quantified by liquid chromatography/mass spectrometry (LC/MS)-based proteomic analysis of CSF from healthy individuals and A-T patients to determine candidate proteins (new biomarkers) which relative expression levels could be used as surrogate marker of disease progression.

DETAILED DESCRIPTION:
Ataxia telangiectasia (A-T) is a devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability, and cancer susceptibility. For clinicians and scientists the underlying mechanism and process of neurodegeneration leading to loss of cerebellar neurons and neurological function is largely unknown. In addition no surrogate marker of neurological degeneration and disease progression exist.

Three major factors may be responsible for progression of neurodegeneration:

1. A-T patients exhibit elevated levels of reactive oxygen species (ROS) and reduced anti-oxidative capacity. It has been proposed that ROS is responsible for destruction of the purkinje cells in the cerebellum.
2. Ongoing low grade inflammation due to immunodeficiency. Elevated serum interleukin-8 (IL-8) levels in patients with A-T are postulated that systemic inflammation may contribute to the disease phenotype. How inflammation and neurodegeneration interact is, however, a matter of ongoing debate.
3. Low levels of growth hormones (GH). Extracerebellar MRI - lesions in A-T go along with deficiency of the GH axis, high Ataxia scores and advanced age.

The aim of the proposal is to investigate oxidative stress, low grade inflammation, tissue breakdown and biomarkers in cerebrospinal fluid (CSF), a fluid that is in direct contact with central nervous system (CNS), of A-T patients.

* To analyse functional gene expression of oxidative stress and low grade inflammation by means of reverse transcriptase-polymerase chain reaction (RT-PCR) and cytometric bead array.
* To characterize the alterations in protein expression related to A-T, a LC/MS-based quantitative proteomic analysis of CSF from control and A-T patients
* To compare alterations in protein expression levels in CSF with MRI findings in different age groups of classical A-T.
* To determine candidate proteins whose relative expression levels could be used as surrogate marker of disease progression?
* To established an analysis system on a basis of multiplex ELISA-technique to evaluate potential candidates/surrogate markers for disease progression in a larger cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aim group: clinically and/or genetically diagnosed Ataxia telangiectasia; Control group: neurologic non-inflammatory disease with an indication for diagnostic or therapeutic lumbar puncture
* age between 2 and 40 years
* written informed consent

Exclusion Criteria:

* fever or clinical signs of an infection
* leucocyte count >12´000/µl and C reactive protein (CrP) >2mg/dl
* chronic diseases with need of immunomodulatory therapies (bronchial asthma, rheumatoid arthritis)
* medication with statins
* other diseases with influence in the immunosystem (i.e. diabetes mellitus, malignoma, renal failure requiring dialysis)

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Concentration of IL-8 and oxidative stress in cerebrospinal fluid | 24 months
  • To analyse functional gene expression of oxidative stress and low grade inflammation by means of RT-PCR and cytometric bead array.

SECONDARY OUTCOMES:
Alterations in protein expression related to A-T | 24 months
  • Alterations in protein expression related to A-T, a LC/MS-based quantitative proteomic analysis of CSF from controls and A-T patients
Number of Participants with Adverse Events | 24 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Alterations in protein expression levels in CSF compared with MRI findings in different age groups of classical A-T. | 24 months
Alterations in protein expression levels in CSF with MRI findings in different age groups of classical A-T. Candidate proteins whose relative expression levels could be used as surrogate marker of disease progression. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospitals, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Hoche F, Seidel K, Theis M, Vlaho S, Schubert R, Zielen S, Kieslich M. Neurodegeneration in ataxia telangiectasia: what is new? What is evident? Neuropediatrics. 2012 Jun;43(3):119-29. doi: 10.1055/s-0032-1313915. Epub 2012 May 21. PMID 22614068
- [Background] Reichenbach J, Schubert R, Schindler D, Muller K, Bohles H, Zielen S. Elevated oxidative stress in patients with ataxia telangiectasia. Antioxid Redox Signal. 2002 Jun;4(3):465-9. doi: 10.1089/15230860260196254. PMID 12215213
- [Background] McGrath-Morrow SA, Collaco JM, Crawford TO, Carson KA, Lefton-Greif MA, Zeitlin P, Lederman HM. Elevated serum IL-8 levels in ataxia telangiectasia. J Pediatr. 2010 Apr;156(4):682-4.e1. doi: 10.1016/j.jpeds.2009.12.007. Epub 2010 Feb 20. PMID 20171651
- [Background] Zielen S, Schubert R. Workshop report: European workshop on ataxia-telangiectasia, Frankfurt, 2011. J Neurogenet. 2011 Oct;25(3):78-81. doi: 10.3109/01677063.2011.592553. Epub 2011 Jul 6. PMID 21732725
- [Background] Dzieciatkowska M, Qi G, You J, Bemis KG, Sahm H, Lederman HM, Crawford TO, Gelbert LM, Rothblum-Oviatt C, Wang M. Proteomic Characterization of Cerebrospinal Fluid from Ataxia-Telangiectasia (A-T) Patients Using a LC/MS-Based Label-Free Protein Quantification Technology. Int J Proteomics. 2011;2011:578903. doi: 10.1155/2011/578903. Epub 2011 Jun 23. PMID 22084690
- See also: Related Info — http://www.info-at.de